CLINICAL TRIAL: NCT04629339
Title: A Phase 2 Study of INCB086550 (Oral PD-L1 Inhibitor) in Participants Who Are Immune Checkpoint Inhibitor-Naïve With Selected Solid Tumors
Brief Title: Study of INCB086550 in Select Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic business decision to terminate the study effective immediately. This is due to a company decision to prioritize another oral PD-L1 inhibitor with a more favorable profile.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 86550-203
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer; Urothelial Cancer; Renal Cell Carcinoma; Hepatocellular Carcinoma; Melanoma
Keywords: checkpoint inhibitor naive; Metastatic; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- INCB086550 (Experimental): INCB086550 will be administered orally twice a day.
  Interventions: Drug: INCB086550

INTERVENTIONS:
Drug: INCB086550 — INCB086550 will be administered orally twice a day.

SUMMARY:
An open-label, nonrandomized study to evaluate the efficacy and safety of INCB086550, a first-in-class oral inhibitor of PD-L1, as initial immune checkpoint inhibitor therapy in participants with select solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Participants with following tumor types : non small cell lung cancer, renal cell carcinoma, urothelial carcinoma, hepatocellular carcinoma and melanoma
* Measurable disease per RECIST v1.1.
* ECOG performance status of 0 to 1 for all tumor types. Urothelial carcinoma allows ECOG of 0 to 2.
* Histologically or cytologically confirmed disease-specific diagnosis as per protocol.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Prior receipt of an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or treatment with an immune modulator (eg, CTLA-4, GITR, LAG3, TIM3, OX40, ICOS, IL2, 4-1BB, CAR-T).
* Receipt of any anticancer therapy or participation in another interventional clinical study.
* Radiotherapy within 14 days of first dose of study treatment.
* Concomitant treatment with moderate and potent CYP3A4/CYP3A5 inhibitors or inducers.
* Toxicity of prior therapy that has not recovered to ≤ Grade 1 or baseline (with the exception of anemia not requiring transfusion support and any grade of alopecia). Endocrinopathy, if well-managed, is not exclusionary and should be discussed with the medical monitor.
* Participant has not recovered adequately from toxicities and/or complications from surgical intervention before starting study drug.
* Participants with laboratory values outside of protocol defined ranges Active malignancy of a type not included in the study population requiring treatment.
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg of prednisone or equivalent).
* Evidence of interstitial lung disease or active, noninfectious pneumonitis.
* Untreated or known active CNS metastases and/or carcinomatous meningitis.
* With the exception of participants with HCC, known active HAV, HBV, or HCV infection, as defined by elevated transaminases with the following serology: positivity for HAV IgM antibody, anti-HCV, anti-HBc IgG or IgM, or HBsAg (in the absence of prior immunization).
* Active infection requiring systemic therapy.
* Receipt of systemic antibiotics within 28 days of first dose of study treatment
* Probiotic usage during screening and throughout the study treatment period.
* Participants who are known to be HIV-positive.
* Participants with impaired cardiac function or clinically significant cardiac disease.
* History or presence of an ECG finding that, in the investigator's opinion, is clinically meaningful.
* Female participant is pregnant or breastfeeding within the projected duration of the study, starting with the screening visit through the 90-day safety follow-up, or male participant is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 100 days after the last dose of study treatment.
* Has received a live vaccine within 90 days of the planned start of study drug.
* Current use of a prohibited medication as described in protocol.
* Life expectancy < 3 months.
* Known hypersensitivity or severe reaction to any component of study drug or formulation components.
* History of organ transplant, including allogeneic stem cell transplantation.
* Inability to swallow tablets or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Bulgaria (4):
  - Complex Oncology Center - Burgas Eood, Burgas
  - Multiprofile Hospital For Active Treatment "Dr. Tota Venkova" Jsc, Gabrovo
  - Complex Onclogy Center Plovdiv Eood, Plovdiv
  - Shatod Dr. Marko - Varna Ltd, Varna
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Complex Oncology Center - Burgas Eood, Farkasgyepű
  - Bacs Kiskun Megyei Oktatokorhaz, Kecskemét
- South Korea (5):
  - The Catholic University of Korea St. Vincent'S Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Chang Gung Memorial Hospital Linkou, Taoyuan, Taiwan
- Ukraine (7):
  - Multifield Clinical Hospital No 4, Dnipro
  - Ci of Healthcare Regional Clinical Specialized Dispensary of the Radiation Protection, Kharkiv
  - Mi Kryviy Rih Center of Dnipropetrovsk Regional Council, Kryvyi Rih
  - Volyn Regional Oncological Dispensary, Lutsk
  - Rmi Sumy Regional Clinical Oncology Dispensary, Sumy
  - Cne Ccch of Uzh Cc Oncological Center, Uzhhorod
  - Medical Clinic Innovacia Llc, Vyshhorod

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 10 study centers in Hungary, Korea, and Ukraine.
Groups:
- NSCLC 400 mg BID: Participants with non-small cell lung cancer (NSCLC) received INCB086550 orally in 28-day cycles at a dose of 400 milligrams (mg) twice daily (BID) for up to 2 years as long as they received benefit and didn't meet any criteria for study withdrawal. Participants who achieved a complete response could have continued to receive INCB086550 for an additional 4 cycles (with a minimum of 1 year of treatment) upon medical monitor consultation.
- UC 400 mg BID: Participants with urothelial carcinoma (UC) received INCB086550 orally in 28-day cycles at a dose of 400 mg BID for up to 2 years as long as they received benefit and didn't meet any criteria for study withdrawal. Participants who achieved a complete response could have continued to receive INCB086550 for an additional 4 cycles (with a minimum of 1 year of treatment) upon medical monitor consultation.
- RCC 400 mg BID: Participants with renal cell carcinoma (RC) received INCB086550 orally in 28-day cycles at a dose of 400 mg BID for up to 2 years as long as they received benefit and didn't meet any criteria for study withdrawal. Participants who achieved a complete response could have continued to receive INCB086550 for an additional 4 cycles (with a minimum of 1 year of treatment) upon medical monitor consultation.
- Melanoma 400 mg BID: Participants with melanoma received INCB086550 orally in 28-day cycles at a dose of 400 mg BID for up to 2 years as long as they received benefit and didn't meet any criteria for study withdrawal. Participants who achieved a complete response could have continued to receive INCB086550 for an additional 4 cycles (with a minimum of 1 year of treatment) upon medical monitor consultation.
- Melanoma 400 mg BID Intermittent Dose: Participants with melanoma received intermittent INCB086550 orally in 28-day cycles at a dose of 400 mg BID. Participants received INCB086550 for 1 week followed by 1 week off for up to 2 years as long as they received benefit and didn't meet any criteria for study withdrawal. Participants who achieved a complete response could have continued to receive INCB086550 for an additional 4 cycles (with a minimum of 1 year of treatment) upon medical monitor consultation.
Period: Overall Study
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose
Started | 1 | 1 | 6 | 7 | 1
Completed | 0 | 0 | 1 | 0 | 1
Not Completed | 1 | 1 | 5 | 7 | 0
Not completed — Death | 1 | 0 | 2 | 2 | 0
Not completed — Disease Progression | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose | Total
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 4 | 5 | 1 | 10
  >=65 years | 1 | 1 | 2 | 2 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 3 | 1 | 8
  Male | 1 | 1 | 2 | 4 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 6 | 7 | 1 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 4 | 7 | 1 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), confirmed by ≥1 repeat assessment ≥28 days later, according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), as determined by the investigator. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 733 days
Population: Full Analysis Set: all study participants who received ≥1 dose of study drug. Participants were analyzed according to the treatment group/dose to which they were assigned. Confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1
percentage of participants | 0.0 [0.0 to 97.5] | 100.0 [2.5 to 100.0] | 0.0 [0.0 to 45.9] | 14.3 [0.4 to 57.9] | 100.0 [2.5 to 100.0]

2. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a best overall response of CR or PR, confirmed by ≥1 repeat assessment ≥28 days later, or stable disease (SD) for ≥12 weeks, by investigator assessment per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. Progressive disease (PD): progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 733 days
Population: Full Analysis Set. Confidence intervals were calculated using the Clopper-Pearson method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1
percentage of participants | 0.0 [0.0 to 97.5] | 100.0 [2.5 to 100.0] | 50.0 [11.8 to 88.2] | 28.6 [3.7 to 71.0] | 100.0 [2.5 to 100.0]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the earliest date of CR or PR, confirmed by ≥1 repeat assessment ≥28 days later, until the earliest date of disease progression by investigator assessment per RECIST v1.1, or death due to any cause, if occurring sooner than progression. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 733 days
Population: Full Analysis Set. Only participants with a CR or PR were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 1
months |  | 3.7 (NA) — Standard deviation cannot be reported for a single participant. |  | 7.4 (NA) — Standard deviation cannot be reported for a single participant. | 23.7 (NA) — Standard deviation cannot be reported for a single participant.

4. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug up to 90 days after the last dose of study drug or until the start of new anticancer therapy, whichever occurred first.
Time Frame: up to 823 days
Population: Safety Evaluable Population: all participants who received ≥1 dose of study drug. Treatment groups for this population were determined according to the actual treatment group/dose the participant received regardless of assigned study drug treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1
Participants | 1 | 1 | 6 | 5 | 1

5. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE
Description: A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug up to 90 days after the last dose of study drug or until the start of new anticancer therapy, whichever occurred first. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events version 5 (CTCAE v5) Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 823 days
Population: Safety Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose
Number analyzed (Participants) | 1 | 1 | 6 | 7 | 1
Participants | 0 | 1 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 90 days after the last dose of study drug or until the start of new anticancer therapy, whichever occurred first (up to approximately 2.5 years)
Description: Adverse events were assessed in members of the Safety Evaluable Population, comprised of all participants who received received ≥1 dose of study drug.
Groups:
- Total: Total
Arm/Group | NSCLC 400 mg BID | UC 400 mg BID | RCC 400 mg BID | Melanoma 400 mg BID | Melanoma 400 mg BID Intermittent Dose | Total
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 2/6 | 2/7 | 0/1 | 5/16
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 2/6 | 0/7 | 0/1 | 3/16
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 6/6 | 5/7 | 1/1 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC 400 mg BID (N=1) | UC 400 mg BID (N=1) | RCC 400 mg BID (N=6) | Melanoma 400 mg BID (N=7) | Melanoma 400 mg BID Intermittent Dose (N=1) | Total (N=16)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NSCLC 400 mg BID (N=1) | UC 400 mg BID (N=1) | RCC 400 mg BID (N=6) | Melanoma 400 mg BID (N=7) | Melanoma 400 mg BID Intermittent Dose (N=1) | Total (N=16)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 2 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Brain compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 3 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligamentum flavum hypertrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 3 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Enrollment in this study was discontinued after INCB086550 program development was terminated by the sponsor due to business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04629339/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04629339/SAP_001.pdf